CLINICAL TRIAL: NCT03799575
Title: Morphology of Internal Limiting Membrane Peeled on Macular Hole Surgery
Brief Title: Internal Limiting Membrane and Macular Hole
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Principal Investigator, Mun Yueh de Faria, MD, Hospital de Santa Maria, Portugal
Other Study IDs: MD26339
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: C11.768.740

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Internal Limiting membrane
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Two samples of ILM per patient are harvested, group A will be immediately fixed and submitted to Optic Microscopy (OM) and Transmission Electron Microscopy (TEM) analysis, and another sample will be incubated in enriched medium 199 (Gibco) for 20 minutes at room temperature, after which it will also be fixed and submitted to OM and TEM analysis.
  Interventions: Behavioral: Transmission Electron Microscopy analysis
- B: Group B sample will be incubated in enriched medium 199 (Gibco) for 20 minutes at room temperature, after which it will also be fixed and submitted to OM and TEM analysis.
  Interventions: Behavioral: Transmission Electron Microscopy analysis

INTERVENTIONS:
Behavioral: Transmission Electron Microscopy analysis — Morphology of two vitreal side of Internal Limiting Membrane in contact

SUMMARY:
Observational study of Internal Limiting Membrane peeled in macular Hole surgery and studied by Transmission electronic Microscopy (TEM) and Optical Coherence Tomography (OCT) findings in closed holes.

DETAILED DESCRIPTION:
A non-randomized prospective study of eyes with MH willing to have surgery at the Department of Ophthalmology of Santa Maria Hospital, Lisbon.

Surgeries are performed under local or general anesthesia, pars plana vitrectomy with internal limiting membrane peeling, fluid gas exchange and face down position.

Two samples of discarded ILM peeled in Macular hole surgery is studied in Laboratory.

Laboratory Analysis Two samples of ILM per patient are harvested, one will be immediately fixed and submitted to Optic Microscopy (OM) and Transmission Electron Microscopy (TEM) analysis, and another sample will be incubated in enriched medium 199 (Gibco) for 20 minutes at room temperature, after which it will also be fixed and submitted to OM and TEM analysis. Both samples from same patient will follow the protocol available at dx.doi.org/10.17504/protocols.io.qjiduke.

Image acquisition Six electron-micrographs will be acquired for each fragment, using a Hitachi H-7000 electron microscope equipped with a megaview III digital camera. Fields of interest will be randomly selected, and acquisition of 15,000x magnification images.

Histology and immunohistochemistry ILM samples will be stained with anti-GFAP antibody (anti-glial fibrillary acidic protein), to detect this protein in glial cells.

Results:

Only successful macular hole closure will be considered, BCVA will be compared before and after surgery and related to OCT findings. ILM findings in TEM analysis will be compared with and without enriched medium.

ELIGIBILITY:
Inclusion Criteria:

* All macular holes were staged based on recent OCT based classification and only full thickness macular hole, grade 2 to 4 IMH are considered for study.

Exclusion Criteria:

* Excluding criteria are maculopathy other than IMH, surgeries of recurrence of IMH, other retinal diseases, or an axial length greater than 26.0 mm. Mean follow-up will be at least 12 months after surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A non-randomized prospective study of eyes with MH willing to have surgery at the Department of Ophthalmology of Santa Maria Hospital, Lisbon.
  Inclusion criteria
  1. Full Thickness Macular Hole
  2. Male or female aged 18 years or older
  3. Visual symptoms due to IMH
  4. Intraocular pressure inferior to 21 mmHG
  5. Signed informed consent form
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-07-02 (Estimated); Study Completion 2019-07-02 (Estimated)

PRIMARY OUTCOMES:
Fibrosis in vitreal sides of Internal Limiting Membranes | 12 months
  Fibrilliary process between two vitreal sides of Internal Limiting Membranes in contact, after incubation in enriched medium

CONTACTS AND LOCATIONS:
Overall Officials: Mun Y Faria, MD, Principal Investigator — Hospital Santa Maria, Centro Hospitalar Universitário Lisboa Norte, 1649-035 Lisboa, PT
Locations (1):
- Hospital Santa Maria, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faria MY, Sousa DC, Almeida BC, Pinto AL, Ferreira NP. Morphology of Peeled Internal Limiting Membrane in Macular Hole Surgery. J Ophthalmol. 2019 May 2;2019:1345683. doi: 10.1155/2019/1345683. eCollection 2019. PMID 31191990